CLINICAL TRIAL: NCT02636114
Title: Effect of Scaling and Root Planing on Serum Renal Function Markers in Systematically Healthy Chronic Periodontitis Subjects - A Control Clinical Trial.
Brief Title: Effect of Scaling and Root Planing on Serum Renal Function Markers in Chronic Periodontitis Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharashtra University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sagar Kadam, Post graduate student, Maharashtra University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MaharashtraUHS
Record Dates: First submitted 2015-12-03; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- scaling and root planing (Active Comparator): this was an international study in which scaling and root planing was done in systemically healthy patients patients with chronic periodontitis
  Interventions: Procedure: scaling and root planing
- control group (No Intervention): Scaling and planing was not done that no intervention is carried out in this group

INTERVENTIONS:
Procedure: scaling and root planing — Scaling and root planing at baseline , checked clinical parameter and serum renal function markers at baseline and 1 month after therapy
  Other Names: Non surgical periodontal therapy
  Arms: scaling and root planing

SUMMARY:
ABSTRACT:-

Introduction:

Chronic periodontitis (CP), the commonest type of periodontal disease, it is an infectious disease resulting in inflammation within of the tissues supporting the teeth, progressive loss of attachment and bone loss. It is closely related to several systemic diseases, such as diabetes and cardiovascular disease. The link between periodontal disease and chronic kidney disease (CKD) may be due to infection and inflammation. The periodontal inflammatory state may increases the chronic inflammation present in CKD, thus decreasing renal function. Periodontal therapy may reduce inflammation and improves endothelial function.

Aim:- To investigate the effect of mechanical non-surgical periodontal therapy on serum renal function markers in systematically healthy CP subjects.

Objectives:- To evaluate the effect of scaling and root planing (SRP) on serum renal function markers such as urea, creatinine, bilurubin in systematically healthy CP patient and to compare the clinical parameters such as Gingival index (GI), Plaque index (PI), Probing depth (PD), Bleeding on probing (BOP), Clinical attachment level (CAL) between test group (TG) & control group (CG).

Materials and Methods: - 51 CP patients; age ranging between 35-60 years was selected. Categorized equally into group I and groups II. Group I was test group (TG) included 25 patients and group II was control group (CG) included 26 patients. The serum levels of renal function markers included Urea, Creatinine, Bilurubin were measured. SRP was done in test group only. All the parameters were checked at baseline and one month after SRP. Comparisons of baseline and value after 1 month among each criterion among each group unpaired-t test and comparisons of two groups for each criterion by paired-t test.

DETAILED DESCRIPTION:
MATERIAL AND METHODS:- A non-surgical interventional clinical study was carried out from January 2015 to March 2015 in 51 patients at the department of Periodontology, Tatyasaheb Kore Dental College & Research Centre, New Pargaon. Prior approval for the study was obtained from the local ethical committee.

Patients with chronic generalized periodontitis [(moderate and severe) according to CDC working group, 2007 criteria]. Age ranging from 35-60 ( mean 45) years, should have at least 20 natural teeth, who have not received periodontal therapy, within preceding six months were included in this study. Tobacco in any form and alcoholics, any other systemic disease which can alter the course of periodontal disease, subjects should have pregnant, women on hormone replacement therapy or hormonal contraceptives, patients taking steroidal or non-steroidal anti-inflammatory drugs (previous 3 months) or antibiotics (previous 6 months), anti-inflammatory drugs and antibiotics in the previous six month and patients with aggressive periodontitis were excluded from this study.

Study was explained, including the benefits, risks and alternative treatments, the patients signed an informed consent form indicating their agreement to participate in the study and each patient was assigned a patient number in ascending order to maintain the masking of evaluators. Eg. First patient is given a number D1, Second D2, and so on.

GROUPS This was a Phase 2 clinical trial with an Interventional model of parallel assignment with two arms. Hence, after screening through inclusion and exclusion criteria patients were divided into two groups, 25 (13 males and 12 females) patients were included in TG and 26 (13 males and 13 females) subjects included in CG.

INTERVENTION:- The study was non-surgical controlled clinical trial. A single study co-ordinator patients into two groups by using Quick Cals, Graph pad software and it has stratified with a 1:1 allocation. SRP had performed for all subjects in TG at baseline by one trained Periodontist under local anaesthesia (if required) using Piezoelectric scaler [Satelec ACTEON P5TM], Hand scalers, Universal curette and Gracey Curette. Clinical and biochemical parameters had recorded by trained examiner in both TG and CG.

BLOOD COLLECTION:- 5 ml of blood was collected from the antecubital fossa by venipuncture using 20-guage needle with 5 ml syringes. Blood samples were left to clot for (1-2) hours, then centrifuged to obtain the serum. Serum was collected in disposable plastic serum containing tube, which was stored at (2-40C) until time of assay. Estimation of levels of urea (by GLDH- urease method), bilirubin total (by Diazo Method), creatinine (modified JAFFE'S method) was done at the baseline and one month in both the groups, at ANANT laboratory, kodoli, Kolhapur (INDIA).

ELIGIBILITY:
Inclusion Criteria:

1. Age group 35-60 years.
2. Subjects should have at least 20 natural teeth.
3. Subjects who have not received periodontal therapy, within preceding six months.
4. Patients with chronic generalized periodontitis (moderate and severe) according to CDC working group, 2007 criteria.

Exclusion Criteria:

1. Tobacco in any form and alcoholics.
2. Any other systemic disease which can alter the course of periodontal disease.
3. Subjects should have pregnant, women on hormone replacement therapy or hormonal contraceptives, patients taking steroidal or non-steroidal anti-inflammatory drugs (previous 3 months) or antibiotics (previous 6 months), anti-inflammatory drugs and antibiotics in the previous six month.
4. Aggressive periodontitis.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
serum creatinine, serum urea, serum bilirubin | 1 month
  to evaluate serum renal markers at baseline and 1 month after scaling and root planing

SECONDARY OUTCOMES:
plaque index | 1 month
  to evaluate plaque index at baseline and 1 month after scaling and root planing
gingival index | 1 month
  to evaluate gingival index at baseline and 1 month after scaling and root planing
pocket depth | 1 month
  to evaluate pocket depth at baseline and 1 month after scaling and root planing
clinical attachment loss | 1 month
  to evaluate clinical attachment loss at baseline and 1 month after scaling and root planing

CONTACTS AND LOCATIONS:
Overall Officials: sagar kadam, MDS, Principal Investigator — muhs
Locations (1):
- Department of Periodontology, Kolhāpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
renal function markers report